CLINICAL TRIAL: NCT04594694
Title: A Phase 2, Double-Blind, Randomized, Parallel Group Study Evaluating the Efficacy, Safety, and Tolerability of Obeticholic Acid Administered in Combination With Bezafibrate in Subjects With Primary Biliary Cholangitis Who Had an Inadequate Response or Who Were Unable to Tolerate Ursodeoxycholic Acid
Brief Title: Study of OCA in Combination With BZF Evaluating Efficacy, Safety, and Tolerability in Participants With PBC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Intercept made a business decision to terminate the study based on FDA's request for voluntary withdrawal of Ocaliva and the issuance of clinical hold on studies under US IND involving OCA.
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 747-213
Record Dates: First submitted 2020-07-14; First posted 2020-10-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary Biliary Cholangitis; Primary Biliary Cirrhosis; PBC; Hepatic Impairment; Cirrhosis; Liver
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fibrosis | interventions — obeticholic acid; Bezafibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Treatment A: BZF 200 milligrams (mg) Immediate release (IR) (Active Comparator): Participants will receive Bezafibrate (BZF) 200 mg IR + OCA Placebo + BZF 400 mg Placebo
  Interventions: Drug: Bezafibrate 200 MG; Drug: OCA Placebo; Drug: Bezafibrate 400 mg Placebo
- Treatment B: BZF 400 mg SR (Active Comparator): Participants will receive BZF 400 mg SR + OCA Placebo + BZF 200 mg Placebo
  Interventions: Drug: OCA Placebo; Drug: Bezafibrate 200 mg Placebo; Drug: Bezafibrate 400 MG
- Treatment C: OCA 5 mg to 10 mg + BZF 200 mg IR (Experimental): Participants will receive OCA 5 mg to 10 mg + BZF 200 mg IR + BZF 400 mg Placebo
  Interventions: Drug: Obeticholic acid; Drug: Bezafibrate 200 MG; Drug: Bezafibrate 400 mg Placebo
- Treatment D: OCA 5 mg to 10 mg + BZF 400 mg SR (Experimental): Participants will receive OCA 5 mg to 10 mg + BZF 400 mg SR + BZF 200 mg Placebo
  Interventions: Drug: Obeticholic acid; Drug: Bezafibrate 200 mg Placebo; Drug: Bezafibrate 400 MG
- Long-term safety extension (LTSE) phase: OCA + BZF (Experimental): Participants will continue the original treatment assignment allocated during the DB Period. The OCA and BZF dose may be optimized based on safety and efficacy during the DB period.
  Interventions: Drug: OCA; Drug: Bezafibrate

INTERVENTIONS:
Drug: Obeticholic acid — 5 mg tablet of OCA once daily titrating up to a maximum of 10 mg OCA once daily
  Arms: Treatment C: OCA 5 mg to 10 mg + BZF 200 mg IR; Treatment D: OCA 5 mg to 10 mg + BZF 400 mg SR
Drug: Bezafibrate 200 MG — 200 mg IR tablet of Bezafibrate once daily for the remainder of the study
  Arms: Treatment A: BZF 200 milligrams (mg) Immediate release (IR); Treatment C: OCA 5 mg to 10 mg + BZF 200 mg IR
Drug: OCA Placebo — One tablet daily for the remainder of the study
  Arms: Treatment A: BZF 200 milligrams (mg) Immediate release (IR); Treatment B: BZF 400 mg SR
Drug: Bezafibrate 200 mg Placebo — One tablet daily for the remainder of the study
  Arms: Treatment B: BZF 400 mg SR; Treatment D: OCA 5 mg to 10 mg + BZF 400 mg SR
Drug: Bezafibrate 400 MG — 400 mg SR tablet of Bezafibrate once daily for the remainder of the study
  Arms: Treatment B: BZF 400 mg SR; Treatment D: OCA 5 mg to 10 mg + BZF 400 mg SR
Drug: Bezafibrate 400 mg Placebo — One tablet daily for the remainder of the study
  Arms: Treatment A: BZF 200 milligrams (mg) Immediate release (IR); Treatment C: OCA 5 mg to 10 mg + BZF 200 mg IR
Drug: OCA — OCA one tablet will be administered.
  Arms: Long-term safety extension (LTSE) phase: OCA + BZF
Drug: Bezafibrate — Bezafibrate one tablet will be administered.
  Arms: Long-term safety extension (LTSE) phase: OCA + BZF

SUMMARY:
Study to evaluate the efficacy, safety, and tolerability of investigational drug obeticholic acid (OCA) in combination with the investigational drug bezafibrate (BZF) in participants with Primary Biliary Cholangitis (PBC).

ELIGIBILITY:
Inclusion Criteria:

* A definite or probable diagnosis of PBC
* Qualifying ALP and/or bilirubin liver biochemistry values
* Taking Ursodeoxycholic Acid (UDCA) for at least 12 months or no UDCA for 3 months before Day 1

Exclusion Criteria:

* History or presence of other concomitant liver diseases
* Clinical complications of PBC
* History or presence of hepatic decompensating events
* Current or history of gallbladder disease
* If female, known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating
* Treatment with commercially available OCA or other farnesoid X receptor (FXR) agonists, or participation in a previous study involving OCA within 3 months before Screening.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Change in Alkaline Phosphatase (ALP) from baseline to Week 12 in the DB Treatment Period | Baseline, Day 1, and Weeks 4, 8, and 12

SECONDARY OUTCOMES:
Response rates of ≥10%, ≥20%, ≥30% and ≥40% reduction, and normalization of biochemical disease marker Alkaline Phosphatase (ALP) | Baseline, Day 1, and Weeks 2, 4, 6, 8, and 12
Number of participants with normalization rates of biochemical disease marker Alanine Aminotransferase (ALT), Gamma-Glutamyl Transpeptidase (GGT), Aspartate Aminotransferase (AST), total and conjugated bilirubin and lipid panel | Baseline, Day 1, and Weeks 2, 4, 6, 8, and 12
Change in GGT from baseline to Week 12 | Baseline, Day 1, and Weeks 4, 8, and 12
Change in ALT from baseline to Week 12 | Baseline, Day 1, and Weeks 4, 8, and 12
Change in AST from baseline to Week 12 | Baseline, Day 1, and Weeks 4, 8, and 12
Change in total and conjugated bilirubin from baseline to Week 12 | Baseline, Day 1, and Weeks 4, 8, and 12
Change in lipid panel from baseline to Week 12 | Baseline, Day 1, and Weeks 4, 8, and 12
Change in 7 alpha (α) hydroxy 4 cholesten-3 one (C4) from baseline to Week 12 | Baseline, Day 1, and Weeks 4, 8, and 12
Change in bile acid from baseline to Week 12 | Baseline, Day 1, and Weeks 4,8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Szczech, Study Director — Intercept Pharmaceuticals, Inc.
Locations (33):
- Australia (2):
  - Flinders Medical Centre, Bedford Park, Perth
  - Royal Adelaide Hospital, Adelaide
- UZ Gasthuisberg, Leuven, Belgium
- Croatia (2):
  - Clinical Hospital Dubrava, Zagreb
  - Zagreb University Hospital Center, Zagreb
- Czechia (3):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Artroscan s.r.o., Gastroenterologicka ambulance, Ostrava
  - Research Site s.r.o., Pilsen
- Tartu University Hospital, Tartu, Estonia
- France (5):
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Groupe Hospitalier Pitié Salpêtrière - Assistance publique - Hôpitaux de Paris, Paris
  - CHU Paris Est - Hopital Saint Antoine, Paris
- Germany (2):
  - Universitatsklinikum Hamburg-Eppendorf UKE, Hamburg
  - Medizinische Hochschule Hannover, Hanover
- Department of Medicine and Research Laboratory of Internal Medicine, University Hospital of Larissa, Larissa, Greece
- Hungary (2):
  - Budai Hepatologiai Centrum (BHC), Budapest
  - DEOEC II. sz. Belgyógyászati Klinika, Debrecen
- Israel (2):
  - Hadassah Ein-Karem Medical Center - Liver unit, Jerusalem
  - Tel Aviv Surasky Medical Center, Tel Aviv
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences, Kauno Klinikos, Kaunas
  - Vlinius University, Vilnius
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Universitetet i Oslo - Akershus Universitetssykehus (AHUS), Loerenskog, Norway
- Narodowy Instytut Onkologii, Klinika Gastroenterologii Onkologicznej, Warsaw, Poland
- South Korea (2):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
- Spain (2):
  - Fundacio Clinic Per La Recerca Biomedica, Barcelona
  - Consorcio Hospital General Universitario, Valencia
- United Kingdom (3):
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Institute of Cellular Medicine, Newcastle University, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Background] Lindor KD, Gershwin ME, Poupon R, Kaplan M, Bergasa NV, Heathcote EJ; American Association for Study of Liver Diseases. Primary biliary cirrhosis. Hepatology. 2009 Jul;50(1):291-308. doi: 10.1002/hep.22906. No abstract available. PMID 19554543
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases. J Hepatol. 2009 Aug;51(2):237-67. doi: 10.1016/j.jhep.2009.04.009. Epub 2009 Jun 6. No abstract available. PMID 19501929